CLINICAL TRIAL: NCT04927598
Title: Predictors and Prognostic Factors of Gullian Barrie Syndrome Outcome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Zayed Saber, principal investigator, Assiut University
Other Study IDs: Gullian Barrie syndrome
Record Dates: First submitted 2021-04-15; First posted 2021-06-16 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Guillain-Barre Syndrome
Keywords: predictors and prognostic factors of outcome
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Plasmapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: plasmapheresis — patients of Gullian Barrie syndrome undergo plasmapharesis

SUMMARY:
This study aims to identify clinical and biological determinants and factors that predict outcome including primary outcome (percentage of changes in clinical scales pre- and after 3 months ) and secondary outcome depending on neurophysiologiacal studies and prognostic factors in individual patients with Guillain-Barre syndrome i individuals managed by plasmapheresis and IVIG immunoglobulin .

This information will be used to understand the diversity in clinical presentation and response to treatment of GBS.

DETAILED DESCRIPTION:
Guillain-Barré syndrome (GBS) is an acute onset, monophasic, immune-mediated peripheral nerve and root disorder (termed polyradiculoneuropathy), GBS has become the most common cause of acute flaccid paralysis worldwide and is a neurological emergency .Guillain-Barré syndrome (GBS) encompasses group of acute immune-mediated disordes restricted to peripheral nerves and roots. Good circumstantial evidence exists for a pathogenic role for molecular mimicry in GBS pathogenesis,especially with its axonal forms, providing insights that could guide future immunotherapy :Intravenous immunoglobulin (IVIg) and plasma exchange (PE) .

Clinical presentation is a sudden onset of rapidly progressive and symmetrical weakness of the limbs, with or without peripheral sensory disturbance, reduction in or loss of tendon reflexes , and cerebrospinal fluid (CSF) analysis showing elevated protein concentrations with a normal white cell count, termed albuminocytologic dissociation, to distinguish it from infections that typically demonstrate elevated protein and white cell counts. The symptoms typically reach maximal severity within four weeks from symptom onset. Most patients generally require hospitalization for treatment, with close cardiopulmonary monitoring performed. Many patients also develop symptoms or signs of autonomic nervous system dysfunction, termed dysautonomia. These commonly consist of sinus tachycardia, arrhythmias,, orthostatic hypotension, increased sweating and bladder and gastrointestinal dysfunction.

Antecedent infections, typically within 4 weeks of neurological symptom onset, commonly occur in GBS patients, resulting in the commonly cited molecular mimicry hypothesis, in which the immune system becomes activated in response to infectious antigen with structural similarity to peripheral nerve myelin or axonal components, with resultant tissue-specific peripheral nerve and nerve root injury in susceptible individuals.

Epidemiological data implies that about two-thirds of GBS adult patients had a prior respiratory or gastrointestinal infection.Pathophysiology and immunopathology of the preceding infections are pathogenically associated with GBS, and may play an essential role in triggering the initial peripheral nerve/ nerve root-specific systemic immune system activation that causes cross-reactive humoral and cellular immune responses with resultant demyelination, axonal injury or both involving peripheral nerves and roots.

Optimal treatment of individual patients may depend on the pathogenesis and clinical severity. Patients with severe forms of GBS may possibly need more intensive treatment to recover. Patients with a milder course that fully recover after standard therapy could suffer from possibly more side effects of more aggressive forms of treatment. This could only be possible if there are prognostic models that accurately predict the clinical course in individual patients. Ideally such models should be based on clinical and biological predictors that are strongly associated with disease course and known as early as possible in the acute phase of illness, when treatment with immunomodulatory therapy is most effective. Prognostic models could help to guide selective trials in specific GBS subtypes. Because of this it will be possible to treat GBS with more effective and more individual therapy

ELIGIBILITY:
Inclusion Criteria:

* Any Age, recent onset of GBS through the first 2 weeks . Gender: Male or Female Inclusion Criteria.

Exclusion Criteria:

* patients with metabolic disorders, others

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Guillian Barre syndrome ( GBS ) is a rare disease , its incidence nearly , 0.8 - 1.8 case / 100000 population ( 16,17) .
  Total coverage of patients with ( GBS ) fitting inclusion criteria and seeking care at Neuro-psychiatric clinics or admitted at Neuro-psychiatry hospital through one year duration about 3 -4 cases per month (36 -38 case per year ) .
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
clinical scales :The GBS Disability Scale | change from baseline scale at 3 months
  the percentage of changes in clinical scales pre- and 3 months after treatment depending on clinical assessment scales : The GBS Disability Scale has six levels: 0 points (healthy), 1 point (minor symptoms and capable of running), 2 points (able to walk 10 m without assistance but unable to run), 3 points (able to walk 10 m across an open space with help), 4 points(bedridden or wheelchair-bound), 5points (requiring assisted ventilation for at least part of the day), and 6 points (dead).
Clinical grading scale MRC ( medial research council sum score ) | change from baseline scale at 3 months
  Clinical grading scale MRC ( medial research council sum score ) from zero ( no power ) up to 60 full power : sum score of muscle power in both upper limbs and lower limbs in points .
ERASMUS GBS respiratory insufficiency score EGRIS : | change from baseline scale at 3 months
  ERASMUS GBS respiratory insufficiency score EGRIS :
  Predict the probability of respiratory insufficiency within the first week of admission, in individual patients with Guillain-Barre . syndrome from zero to 7 points score : 0 point ( no affection ) , 7 point ( severe affection )
Erasmus GBS Outcome Score (EGOS) | change from baseline scale at 3 months
  Erasmus GBS Outcome Score (EGOS) is a prognostic model based on age, diarrhea, and GBS disability score at 2 weeks after hospital admission that accurately predicts the chance of being able to walk independently at 3 months
overall neuropathy limitations scale ONLS . | change from baseline scale at 3 months
  it is modified disability sum score : sum of arm grade and leg grade limitation score ; arm grade from zero point ( less limitation ) to 5 points ( most limitation ) and leg grade from zero point ( less limitation) to 7 points (more limitation)

SECONDARY OUTCOMES:
comparison between pre and post neurophysiological studies | change from baseline scale at 3 months
  neurophysiological study pre- and after 3 months change of degree of affection and improvement in latency in nerve conduction m/ sec. amplitude m/v , velocity of nerve /s conduction and F-wave of both upper limbs and lower limbs

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] van Doorn PA, Ruts L, Jacobs BC. Clinical features, pathogenesis, and treatment of Guillain-Barre syndrome. Lancet Neurol. 2008 Oct;7(10):939-50. doi: 10.1016/S1474-4422(08)70215-1. PMID 18848313
- [Background] Raphael JC, Chevret S, Hughes RA, Annane D. Plasma exchange for Guillain-Barre syndrome. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD001798. doi: 10.1002/14651858.CD001798.pub2. PMID 22786475
- [Background] Fokke C, van den Berg B, Drenthen J, Walgaard C, van Doorn PA, Jacobs BC. Diagnosis of Guillain-Barre syndrome and validation of Brighton criteria. Brain. 2014 Jan;137(Pt 1):33-43. doi: 10.1093/brain/awt285. Epub 2013 Oct 26. PMID 24163275
- [Background] van Doorn PA. Diagnosis, treatment and prognosis of Guillain-Barre syndrome (GBS). Presse Med. 2013 Jun;42(6 Pt 2):e193-201. doi: 10.1016/j.lpm.2013.02.328. Epub 2013 Apr 28. PMID 23628447
- [Background] van Nes SI, Vanhoutte EK, van Doorn PA, Hermans M, Bakkers M, Kuitwaard K, Faber CG, Merkies IS. Rasch-built Overall Disability Scale (R-ODS) for immune-mediated peripheral neuropathies. Neurology. 2011 Jan 25;76(4):337-45. doi: 10.1212/WNL.0b013e318208824b. PMID 21263135
- [Background] Mori M, Kuwabara S, Fukutake T, Hattori T. Intravenous immunoglobulin therapy for Miller Fisher syndrome. Neurology. 2007 Apr 3;68(14):1144-6. doi: 10.1212/01.wnl.0000258673.31824.61. PMID 17404197
- [Background] Kalita J, Misra UK, Goyal G, Das M. Guillain-Barre syndrome: subtypes and predictors of outcome from India. J Peripher Nerv Syst. 2014 Mar;19(1):36-43. doi: 10.1111/jns5.12050. PMID 24456386
- [Background] Dornonville de la Cour C, Jakobsen J. Residual neuropathy in long-term population-based follow-up of Guillain-Barre syndrome. Neurology. 2005 Jan 25;64(2):246-53. doi: 10.1212/01.WNL.0000149521.65474.83. PMID 15668421
- [Background] van Koningsveld R, Steyerberg EW, Hughes RA, Swan AV, van Doorn PA, Jacobs BC. A clinical prognostic scoring system for Guillain-Barre syndrome. Lancet Neurol. 2007 Jul;6(7):589-94. doi: 10.1016/S1474-4422(07)70130-8. PMID 17537676
- [Background] Walgaard C, Lingsma HF, Ruts L, van Doorn PA, Steyerberg EW, Jacobs BC. Early recognition of poor prognosis in Guillain-Barre syndrome. Neurology. 2011 Mar 15;76(11):968-75. doi: 10.1212/WNL.0b013e3182104407. PMID 21403108
- [Derived] Khedr EM, Shehab MM, Mohamed MZ, Mohamed KO. Early electrophysiological study variants and their relationship with clinical presentation and outcomes of patients with Guillain-Barre syndrome. Sci Rep. 2023 Aug 26;13(1):14000. doi: 10.1038/s41598-023-41072-x. PMID 37634022